CLINICAL TRIAL: NCT04912297
Title: Persistence of Humoral Immunity to Serotype 19A Streptococcus Pneumoniae in Children Vaccinated With the 10-valent Pneumococcal Conjugate Vaccine in Finland
Brief Title: Immunity to Serotype 19A Streptococcus Pneumoniae in Children Vaccinated With PCV10
Status: Completed | Type: Observational
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Turku University Hospital (Other Government); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: THL/1019/6.00.00/2017
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Pneumococcal Infections
Keywords: Streptococcus pneumoniae; antibody
MeSH Terms: conditions — Pneumococcal Infections | interventions — 10-valent pneumococcal conjugate vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Serum samples collected at 13 months, 2 years or 3 years from children vaccinated with PCV10 with 2+1 or 3+1 schedule
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- PCV10 2+1 schedule: Ten-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10; GlaxoSmithKline) administered with a 2+1 schedule (two vaccinations with minimum 8-week intervals followed by a booster dose at least 4 months after the last primary dose).
  Interventions: Biological: 10-valent pneumococcal conjugate vaccine, PCV10
- PCV10 3+1 schedule: Ten-valent pneumococcal Haemophilus influenzae protein D conjugate vaccine (PHiD-CV10; GlaxoSmithKline) administered with a 3+1 schedule (three vaccinations with minimum 4-week intervals, followed by a booster dose at least 4 months after the last primary dose).
  Interventions: Biological: 10-valent pneumococcal conjugate vaccine, PCV10

INTERVENTIONS:
Biological: 10-valent pneumococcal conjugate vaccine, PCV10 — 10-valent pneumococcal conjugate vaccine, PCV10

SUMMARY:
The aim of the study are to assess the persistence of immunity against vaccine serotypes (VSTs) and vaccine-related serotypes in PCV10 vaccinated children in Finland.

DETAILED DESCRIPTION:
The primary objective is to evaluate the long-term persistence of humoral immunity to vaccine-related pneumococcal serotypes after vaccination with PCV10.

ELIGIBILITY:
Inclusion Criteria:

* Completed PCV10 vaccination with 3 or 4 doses (2+1 or 3+1 schedule) before blood sampling at age of 13 months
* Age at sample collection 13 months, 2 years or 3 years
* PCV10 vaccination received 2-6 weeks before sample collection at the age of 1 year
* Informed consent obtained covering the planned analyses

Exclusion Criteria:

* PCV13 or PPV23 dose received
* Informed consent withdrawn

Ages: 13 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born in 2008-2010 in the Hospital District of Southwest Finland. These children participated in the Finnish Invasive Pneumococcal Disease (FinIP) Vaccine Trial before introduction of PCV10 into the national immunization program in 2010. Serum samples from the children were collected in The Steps to the Healthy Development and Well-being of Children (STEPS) Study at the ages of 13 months, 2 years and 3 years.
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2009-11-12 (Actual); Primary Completion 2013-05-07 (Actual); Study Completion 2013-05-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arto Palmu, MD, PhD, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- Finnish Institute for Health and Welfare, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PCV10 2+1 Schedule | PCV10 3+1 Schedule
Started | 99 | 87
Completed | 68 | 54
Not Completed | 31 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCV10 2+1 Schedule | PCV10 3+1 Schedule | Total
Number analyzed (Participants) | 68 | 54 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 68 | 54 | 122
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 58
  Male | 35 | 29 | 64
Region of Enrollment [Number; unit: participants]
  Finland | 68 | 54 | 122

OUTCOME MEASURES:

1. Primary Outcome: Persistence of Humoral Immunity Following PCV10 Vaccination
Description: Persistence of humoral immunity to vaccine- and vaccine-related pneumococcal serotypes after vaccination with PCV10. The serotype 19A specific geometric mean IgG antibody concentrations are reported as micrograms per ml with 95% confidence intervals.
Time Frame: Two years following last PCV10 vaccination
Population: IgG concentrations to serotype 19A at two years following last PCV vaccination in subjects vaccinated with PCV10 with a 2+1 or 3+1 schedule
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per ml
Arm/Group | PCV10 2+1 Schedule | PCV10 3+1 Schedule
Number analyzed (Participants) | 68 | 54
micrograms per ml | 0.32 [0.22 to 0.48] | 0.35 [0.23 to 0.53]

ADVERSE EVENTS:
Arm/Group | PCV10 2+1 Schedule | PCV10 3+1 Schedule
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/54
Other Adverse Events (participants affected / at risk) | 0/68 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes